CLINICAL TRIAL: NCT05140889
Title: Integrating Deep Learning CT-scan Model, Biological and Clinical Variables to Predict Severity of Asthma in Children
Acronym: BREATHE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Istituto per la Ricerca e l'Innovazione Biomedica (Other); Università Ca' Foscari Venezia (Unknown)
Responsible Party: Principal Investigator, Amelia Licari, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 08073521
Record Dates: First submitted 2021-10-13; First posted 2021-12-02 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children
Keywords: Asthma; Children; Severe Asthma; Artificial Intelligence; Deep Learning; Computed Tomography
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children with severe asthma
- Group 2: Children who undergo chest CT scan for other reasons than asthma

SUMMARY:
Artificial intelligence (AI) offers substantial opportunities for healthcare, supporting better diagnosis, treatment, prevention and personalized care. Analysis of health images is one of the most promising fields for applying AI in healthcare, contributing to better prediction, diagnosis and treatment of diseases.

Deep learning (DL) is currently one of the most powerful machine learning techniques. DL algorithms are able to learn from raw (or with little pre-processing) input data and build by themselves sophisticated abstract feature representations (useful patterns) that enable very accurate task decision making. Recently, DL has shown promising results in assisting lung disease analysis using computed tomography (CT) images.

Current severe asthma guidelines recommend high-resolution and multidetector CT as a tool for disease evaluation. CT scans contain prognostic information, as the presence of bronchial wall thickening, air trapping, bronchial luminal narrowing, and bronchiectasis are associated with longer disease duration and disease severity in adults. Only a small number of studies have reported chest CT findings in children with severe asthma, and their relationship to clinical and pathobiological parameters yielded inconsistent results. Thus, to which extent CT scans add prognostic information beyond what can be inferred from clinical and biological data is still unresolved in children.

The project is expected to build an DL-severity score to prognoses severe evolution for children with asthma, using a DL model to capture CT scan prognosis information.

DETAILED DESCRIPTION:
The aims of this project are:

* to build a large database of clinical, biological and radiological data collected from pediatric patients with severe asthma;
* to design and train a forecaster model based on DL techniques to predict asthma severity in children;
* to estimate transition probabilities between asthma severity levels using a multi-state Markov model taking into account qualitative and quantitative information obtained from CT imaging.

Our evaluation of DL-severity and existing clinical scores in childhood asthma is expected to reveal that emerging methodologies assisted by DL techniques can provide accurate severity predictions, when compared with existing clinical scores. Such an accurate prediction model would allow pediatricians to identify features that are the most indicative of severity and progression of asthma and would be employed to formulate intervention strategies and early medical attention for children.

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years
* confirmed diagnosis of severe asthma according to ERS/ATS guidelines

Exclusion Criteria:

* other diseases that may mimic asthma according to ERS/ATS guidelines (i.e., cystic fibrosis, primary ciliary dyskinesia, tracheobronchomalacia, etc)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible participants will be identified among children referred to our Pediatric Clinic for severe asthma by their general practitioner or by their primary care pediatrician.
  Children who undergo chest CT scan for other reasons than asthma will be selected as controls.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prediction of asthma severity in children | 3 years
  To build a severity score to prognoses evolution for children with asthma, using a deep-learning model to capture CT scan prognosis information and integrate with clinical and laboratory data obtained from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Licari, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No